CLINICAL TRIAL: NCT03452553
Title: A Prospective, US Multicenter Open Label Study in the Treatment of Hepatocellular Carcinoma (HCC) With a Radiopaque (RO) Bead (LC Bead LUMI™) Loaded With Doxorubicin
Brief Title: Study in the Treatment of HCC With a Radiopaque (RO) Bead (LC Bead LUMI™) Loaded With Doxorubicin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: CMS disapproval, no alternative for sites/patient, risk of financial burden.
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatabilities UK Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTG004387-01
Record Dates: First submitted 2018-02-12; First posted 2018-03-02 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Liver Cancer; Hepatocellular Carcinoma (HCC); Trans Arterial Chemo Embolization (TACE); Drug Eluting Beads (DEB); Doxorubicin (DOX)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Open Label Treatment (Experimental): Chemoembolization using LC Bead LUMI™ (Radiopaque (RO) Bead) loaded with doxorubicin
  Interventions: Device: LC Bead LUMI™ (Radiopaque (RO) Bead) loaded with doxorubicin

INTERVENTIONS:
Device: LC Bead LUMI™ (Radiopaque (RO) Bead) loaded with doxorubicin — Drug Eluting Beads loaded with chemotherapy

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common type of primary liver cancer. This type of cancer may be "hypervascular". Hypervascular means there is an increased number or concentration of blood vessels. These blood vessels get their blood supply from the hepatic artery, while the non-tumor liver tissue gets blood supply from the portal vein. Therefore, blockage of the hepatic artery to cut off the blood supply to the tumor is possible without affecting the normal liver.

This research protocol will study chemoembolization using radiopaque beads loaded with a chemotherapy drug called doxorubicin. Chemoembolization is a procedure in which the blood supply to a tumor is blocked after anticancer drugs are given in blood vessels near the tumor. In this study, the anticancer drug, doxorubicin, is attached to small beads that are injected into an artery that feeds the tumor. The radiopaque beads (RO beads) are visible on imagining scans (X-rays) so that the Interventional Radiologist performing the chemoembolization procedure can see the location of the beads in the tumor during and after the procedure. The visibility of the beads allows the interventional radiologist to confirm where the beads loaded with doxorubicin have been delivered in the tumor; this in theory could help to improve the efficiency of embolization and plan the next course of treatment. In addition to the embolization, the beads elute a sustained dose of doxorubicin locally to the tumor site as a second effect.

DETAILED DESCRIPTION:
The usual treatment for HCC is to perform a procedure to the tumor known as Transarterial Chemo-Embolization (TACE). TACE has been approved and used worldwide for over 10 years.

Transarterial means that the treatment is delivered using a catheter inserted into the hepatic artery. Embolization is a treatment that blocks or slows down the blood supply to tissues. This procedure is performed to block the flow of blood to a tumor, so the cancer cells die because the oxygen supply is interrupted. When the material used to block the blood supply also delivers a chemotherapy drug to the tumor, it is called chemoembolization. The most commonly used material for chemoembolization are drug-eluting beads (DEBs) that are loaded with a chemotherapy drug (doxorubicin). These beads are not visible, during the procedure, on the imaging (scanner, ultrasonography or MRI) while injected into the tumor. The consequences of the blood flow interruption are visible on imaging (CT, MRI) in the weeks following treatment (tissue infarction/tumor necrosis).

This study uses the LC Bead LUMI™ radiopaque beads (RO beads). The difference is that RO Beads are visible with X-Ray imaging (scanner, fluoroscopy). This is important because it means that the Interventional Radiologist is able to verify, during the procedure, where the beads have been delivered to the tumor. The Interventional Radiologist will identify the blood supply to the tumor, and then inject the LC Bead LUMI™ loaded with doxorubicin and a compatible contrast agent into the blood vessels that supply the liver tumor. These RO beads block the blood vessel, starve the tumor of nutrients and deliver a slow release of the doxorubicin.

Many of the tests, investigations and procedures that will be requested as a part of the study may be the same as what is routinely done in the diagnosis and treatment of HCC. These tests will be used to determine if you are eligible to participate in this study and receive the LC Bead LUMI™ loaded with doxorubicin. Some of the study assessments are done to evaluate the safety and efficacy of the treatment procedure and others will be done for research purposes.

During the study, the tests and evaluations will be scheduled with normally occurring appointments, when possible; to reduce the number of visits the patient needs to make to the study center. Study visits for tumor response evaluation occur at one month after the first treatment then every 3 months for 2 years then every 6 months.

The information obtained during your visits will help your study doctor determine what choices you have for the next best course of action in treating your cancer. Options may include; repeat the study treatment, propose another alternative treatment or to continue the follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with HCC, diagnosed by at least one of the following:

   1. Imaging according to the American Association for the Study of Liver Disease (AASLD) guidelines
   2. Histology
2. Adults (18 years of age or older)
3. Tumor not suitable for resection, ablation or transplantation at the time of study entry
4. Patient is a candidate for TACE after multidisciplinary team (MDT) decision
5. HCC Barcelona Clinic Liver Cancer (BCLC) B or BCLC A not eligible for or refuses curative treatment, or BCLC C (Performance Status 1 only)
6. At least one measurable disease according to mRECIST
7. Preserved liver function (Child Pugh Score A and B7)
8. Performance Status: Eastern Cooperative Oncology Group score of 0 or 1 or Karnofsky Performance Status 80 -100 at study entry
9. TACE of all lesions can be achieved within a single cycle (2 sessions in 21 days +/- 7 days for the first cycle only)
10. Life expectancy of at least 6 months at study entry
11. Women and men of child bearing potential must agree to use adequate contraception prior, during and post therapy according to the standard instructions at the study site
12. Negative serum or urine pregnancy test at study entry for woman of childbearing potential according to institutional policy
13. Patient is willing and able to provide written signed and dated informed consent

Exclusion Criteria:

1. Extrahepatic metastases
2. Portal vein tumor thrombosis (any type I to IV, refer to appendix 12.6)
3. Patient on waiting list for transplantation
4. Hematology:

   1. Hemoglobin <9g/dL, or
   2. White Blood Cell (WBC) <2,500 cells/mm3, or
   3. Absolute Neutrophil Count (ANC) <1,500 cells/mm3, or
   4. Platelets <50,000/mm3, or
   5. International Normalized Ratio (INR) > 1.8
5. Renal

   1. Glomerular Filtration Rate (GFR) <30 mL/min/1.73m2
   2. Creatinine >2 mg/dL
6. Hepatic

   1. Any single tumor nodule > 7cm (Multiple lesions can be included but not one >7cm)
   2. Estimated tumor burden >50%
   3. Clinically detectable ascites on physical exam (ascites detected by imaging only and is deemed not clinically significant is acceptable)
   4. Bleeding diathesis; history of hemorrhage / bleeding events
   5. Variceal bleeding of grade 3 or worse within 3 months of study entry
   6. Bilirubin >3mg/dL,
   7. Significant impairment of liver function tests defined as AST/ALT >5X Upper Limit Normal or 250 units/L
   8. Albumin <30g/L
7. Cardiovascular

   a. Significant cardiovascular disease; e.g., myocardial infarction within 6 months of inclusion, chronic heart failure (New York Heart Association class III or IV), Left Ventricular Ejection Fraction <50%, unstable coronary artery disease
8. Other serious concurrent medical conditions

   1. Previous malignancy other than carcinoma in situ of the skin, the cervix or uterus within 5 years prior to inclusion
   2. HIV, congenital immune defect, any immunosuppressive therapy for autoimmune disease (rheumatoid arthritis) or inflammatory bowel disease
   3. History of organ transplant
   4. Serious or chronic infection (Active, clinically severe bacteria or fungal infection of >grade 2 NCI-CTCAE_ v4.0)
   5. In case of Hepatitis B or C, viral disease must be under control (antiviral treatment not needed or completed or if hepatitis B with no interaction with cancer treatment).
   6. Other uncontrolled intercurrent underlying medical condition that in judgement of the investigator could impact the ability of the subject to participate in the trial
9. Prior or concurrent cancer therapy

   1. Target lesions previously treated by a loco regional therapy (TACE, Y90, RFA, MWA, PEI, SBRT)
   2. Any systemic treatment within the past 3 months or any plan to administer systemic treatments during the study
   3. Endocrine therapy - any prior hormonal therapy for HCC
   4. Radiotherapy - any prior radiotherapy for HCC or any concurrent anticancer radiotherapy
   5. Surgery - major surgery/laparoscopy within 30 days before screening
   6. Investigational therapy - Patients who have participated in another clinical study within 12 weeks prior to the Screening/Baseline visit
   7. TACE therapy - Prior TACE on the same lesions
10. Performance Status: ECOG ≥ 2 or KPS < 80 at study entry
11. Contraindication for both enhanced Magnetic Resonance Imaging (MRI) and Computerized Tomography (CT) imaging (according to patient characteristics and investigator decision).
12. Any condition that would result in biliary ductal colonization including Whipple procedure, biliary stenting, a sphincterotomy within 3 month, hepatojejunostomy, etc.
13. Mental conditions rendering the subject incapable to understand the nature, scope, and consequences of the trial
14. Any absolute contra-indication to TACE, contraindication to angiography
15. Any absolute contra-indication to doxorubicin according to its label
16. Contraindication or known allergic reactions to contrast media agents, Radiopaque Beads or with known sensitivity to iodine/iodine containing substances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Time to progression (TTP) | 12 months
  Time when progression is first observed at a tumor assessment according to mRECIST evaluated by CT scan or MRI.

SECONDARY OUTCOMES:
Safety: Adverse Events (AE) and Serious Adverse Events (SAE) | Assessed at 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months post first treatment
  The incidence of treatment emergent AE's and SAE's will be summarized according to the standardized grading criteria (NCI CTCAEv4.0).
Objective Response Rate (ORR) and Disease Control Rate (DCR) | Assessed at 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months post first treatment
  ORR is defined as a complete response or partial response, DCR is defined as a complete response, partial response or stable disease, according to mRECIST evaluated by CT or MRI.
Time to local progression (TTLP) | Assessed at 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months post first treatment
  Progression of Target Lesion response according to mRECIST evaluated by CT or MRI.
Overall survival (OS) | Assessed at 1, 3, 6, 9, 12, 15, 18, 21, 24, 30 and 36 months
  Assessment of overall survival for all subjects until death any cause
Physician rating of the handling and visibility of LC Bead LUMI™. | Intra and post intervention at Day 1, and 6 and 12 months post first treatment.
  Investigator rating of deposition and handling of the study device

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolondi L, Burroughs A, Dufour JF, Galle PR, Mazzaferro V, Piscaglia F, Raoul JL, Sangro B. Heterogeneity of patients with intermediate (BCLC B) Hepatocellular Carcinoma: proposal for a subclassification to facilitate treatment decisions. Semin Liver Dis. 2012 Nov;32(4):348-59. doi: 10.1055/s-0032-1329906. Epub 2013 Feb 8. PMID 23397536
- [Background] Bosetti C, Levi F, Boffetta P, Lucchini F, Negri E, La Vecchia C. Trends in mortality from hepatocellular carcinoma in Europe, 1980-2004. Hepatology. 2008 Jul;48(1):137-45. doi: 10.1002/hep.22312. PMID 18537177
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] Chan SL, Chong CC, Chan AW, Poon DM, Chok KS. Management of hepatocellular carcinoma with portal vein tumor thrombosis: Review and update at 2016. World J Gastroenterol. 2016 Aug 28;22(32):7289-300. doi: 10.3748/wjg.v22.i32.7289. PMID 27621575
- [Background] El-Serag HB. Epidemiology of viral hepatitis and hepatocellular carcinoma. Gastroenterology. 2012 May;142(6):1264-1273.e1. doi: 10.1053/j.gastro.2011.12.061. PMID 22537432
- [Background] European Association for Study of Liver; European Organisation for Research and Treatment of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. Eur J Cancer. 2012 Mar;48(5):599-641. doi: 10.1016/j.ejca.2011.12.021. No abstract available. PMID 22424278
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Johnson CG, Tang Y, Beck A, Dreher MR, Woods DL, Negussie AH, Donahue D, Levy EB, Willis SL, Lewis AL, Wood BJ, Sharma KV. Preparation of Radiopaque Drug-Eluting Beads for Transcatheter Chemoembolization. J Vasc Interv Radiol. 2016 Jan;27(1):117-126.e3. doi: 10.1016/j.jvir.2015.09.011. Epub 2015 Nov 6. PMID 26549370
- [Background] Hashim D, Boffetta P, La Vecchia C, Rota M, Bertuccio P, Malvezzi M, Negri E. The global decrease in cancer mortality: trends and disparities. Ann Oncol. 2016 May;27(5):926-33. doi: 10.1093/annonc/mdw027. Epub 2016 Jan 22. PMID 26802157
- [Background] Idee JM, Guiu B. Use of Lipiodol as a drug-delivery system for transcatheter arterial chemoembolization of hepatocellular carcinoma: a review. Crit Rev Oncol Hematol. 2013 Dec;88(3):530-49. doi: 10.1016/j.critrevonc.2013.07.003. Epub 2013 Aug 6. PMID 23921081
- [Background] Lencioni R, de Baere T, Burrel M, Caridi JG, Lammer J, Malagari K, Martin RC, O'Grady E, Real MI, Vogl TJ, Watkinson A, Geschwind JF. Transcatheter treatment of hepatocellular carcinoma with Doxorubicin-loaded DC Bead (DEBDOX): technical recommendations. Cardiovasc Intervent Radiol. 2012 Oct;35(5):980-5. doi: 10.1007/s00270-011-0287-7. Epub 2011 Oct 19. PMID 22009576
- [Background] Levy EB, Krishnasamy VP, Lewis AL, Willis S, Macfarlane C, Anderson V, van der Bom IM, Radaelli A, Dreher MR, Sharma KV, Negussie A, Mikhail AS, Geschwind JF, Wood BJ. First Human Experience with Directly Image-able Iodinated Embolization Microbeads. Cardiovasc Intervent Radiol. 2016 Aug;39(8):1177-86. doi: 10.1007/s00270-016-1364-8. Epub 2016 May 20. PMID 27206503
- [Background] McGlynn KA, Petrick JL, London WT. Global epidemiology of hepatocellular carcinoma: an emphasis on demographic and regional variability. Clin Liver Dis. 2015 May;19(2):223-38. doi: 10.1016/j.cld.2015.01.001. Epub 2015 Feb 26. PMID 25921660
- [Background] Pons F, Varela M, Llovet JM. Staging systems in hepatocellular carcinoma. HPB (Oxford). 2005;7(1):35-41. doi: 10.1080/13651820410024058. PMID 18333159
- [Background] Ryerson AB, Eheman CR, Altekruse SF, Ward JW, Jemal A, Sherman RL, Henley SJ, Holtzman D, Lake A, Noone AM, Anderson RN, Ma J, Ly KN, Cronin KA, Penberthy L, Kohler BA. Annual Report to the Nation on the Status of Cancer, 1975-2012, featuring the increasing incidence of liver cancer. Cancer. 2016 May 1;122(9):1312-37. doi: 10.1002/cncr.29936. Epub 2016 Mar 9. PMID 26959385
- [Background] Weinmann A, Koch S, Sprinzl M, Kloeckner R, Schulze-Bergkamen H, Duber C, Lang H, Otto G, Worns MA, Galle PR. Survival analysis of proposed BCLC-B subgroups in hepatocellular carcinoma patients. Liver Int. 2015 Feb;35(2):591-600. doi: 10.1111/liv.12696. Epub 2014 Oct 31. PMID 25290314
- See also: Sponsor Website — http://www.btgplc.com